CLINICAL TRIAL: NCT03396406
Title: Comparison of Extended Duration Pulsed Radiofrequency Plus Low Temperature Thermal Radiofrequency With Thermal Radiofrequency Alone in Treatment of Recurrent Trigeminal Neuralgia
Brief Title: Treatment of Recurrent Trigeminal Neuralgia by Using Extended Duration of Pulsed Radiofrequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Assistant professor of Anesthesia and Intensive care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB0000871244
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Trigeminal Neuralgia
Keywords: trigeminal neuralgia, radiofrequency
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Pulsed Radiofrequency Treatment; Electrocoagulation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCRF group (Experimental): received Pulsed radiofrequency (PRF) at 42°C for 8 minutes followed by CRF at 60°C for 270s
  Interventions: Device: Pulsed radiofrequency (PRF)
- CRF group (Experimental): received sole thermocoagulation at 70°C for 270 s
  Interventions: Device: thermocoagulation

INTERVENTIONS:
Device: Pulsed radiofrequency (PRF) — received PRF at 42°C for 8 minutes followed by CRF at 60°C for 270s
  Arms: PCRF group
Device: thermocoagulation — received sole CRF at 70°C for 270 s
  Arms: CRF group

SUMMARY:
Forty patients with history of recurrent TN were recruited in Assiut University Hospitals, Pain Unit from 2012 to 2017. Before the study, all patients were given adequate and informative data about the nature of the study, interventional procedure and its possible complications, and a well-informed written consent was obtained from each patients.

DETAILED DESCRIPTION:
All interventions were done in a specialized well-equipped unit at Assiut University hospital and continuous hemodynamic monitoring with pulse oximetry, blood pressure and ECG applied for each patient. Light sedation by using midazolam 5mg bolus. In a supine position with slightly extended head and under fluoroscopic control, C arm rotated caudo-cranially and ipsilateraly to produce an oblique submental view and visualize foramen ovale beside the ramus of the mandible. The point of entry varied according to the affected branch, but it ranged from 0.5-1.5 cm from the corner of the mouth. The point of entry cleaned by aseptic solution and anaesthetized with 1% of Lidocaine. C arm has been rotated laterally to confirm the depth of penetration once the needle entered into Meckel's cavity. RF electrode (22-G, 10 cm needle, with a curved 5 mm active tip, Neurotherm 1100) was used and the exact position of the needle confirmed by sensory stimulation, motor stimulation and negative aspiration as the following criteria:-

1. Sensory stimulation (50 Hz) threshold between 0.1-0.3 V which made paresthesia and/ or tingling in the affected painful area. Patient was awake to respond to the sensory stimulation
2. Motor stimulation at 2Hz with 0.1-1.5V caused muscle contraction of the lower mandible.

After confirming the position of the RF electrode, each patient received 0.5 ml of 1% of Lidocaine to avoid discomfort during treatment. Then the type of intervention determined by the person who was responsible for randomisation process and who did not involve in assessing eligibility or interventional technique and divided into:-

* Group A: pulsed radiofrequency was applied for 4 cycles of 120 seconds ( 8 minutes in total) at 45 V and temperature was set at 42 C. then conventional radiofrequency thermal lesion was applied for 3 cycles of 90 seconds at 60 c.
* Group B: thermal energy was applied gradually for 3 cycles of 90 seconds at 70 C.

ELIGIBILITY:
Inclusion Criteria:

* • Patient with severe, recurrent TN for more than 6 months, non-satisfactory pain relief with medical treatment or/and intolerable to medical drugs

  * Age more than 18 years old
  * Pain score ≥ 7
  * Patient consent to participate

Exclusion Criteria:

* • Known concurrent neurological or neurodegenerative diseases such as multiple sclerosis, and myasthenia gravis

  * Breast feeding or pregnant women
  * Advanced malignancy or brain stem tumors
  * Coagulopathy or patients on anticoagulant medications
  * Allergy/ sensitivity to Lidocaine anesthetic or/and non- ionic contrast media
  * Presence of Progressive Motor or sensory deficit in the distribution of trigeminal nerve
  * Active psychological or mental diseases
  * Uncontrolled medical or respiratory conditions
  * Patients who are unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Visual analog pain score | one month
  The response for interventional treatment was evaluated in subsequent visits at pain clinic or by telephone
Visual analog pain score | 6 months
  The response for interventional treatment was evaluated in subsequent visits at pain clinic or by telephone
Visual analog pain score | one year
  The response for interventional treatment was evaluated in subsequent visits at pain clinic or by telephone
Visual analog pain score | 2 years
  The response for interventional treatment was evaluated in subsequent visits at pain clinic or by telephone

SECONDARY OUTCOMES:
change in medical treatment | 2 years
  need for tricyclic antidepressant

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrady S Ibrahim, M.D., Principal Investigator — Assiut university faculty of medicine
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elias WJ, Burchiel KJ. Microvascular decompression. Clin J Pain. 2002 Jan-Feb;18(1):35-41. doi: 10.1097/00002508-200201000-00006. PMID 11803301
- [Derived] Abdel-Rahman KA, Elawamy AM, Mostafa MF, Hasan WS, Herdan R, Osman NM, Ibrahim AS, Aly MG, Ali AS, Abodahab GM. Combined pulsed and thermal radiofrequency versus thermal radiofrequency alone in the treatment of recurrent trigeminal neuralgia after microvascular decompression: A double blinded comparative study. Eur J Pain. 2020 Feb;24(2):338-345. doi: 10.1002/ejp.1489. Epub 2019 Oct 16. PMID 31571339